CLINICAL TRIAL: NCT07035288
Title: Electroanatomical Mapping Versus Fluoroscopy Based Pulmonary Vein Isolation by Means of PulseSelect Catheter in Patients With Atrial Fibrillation
Brief Title: PulseSelect Based Pulmonary Vein Isolation and Ablation in Patients With Atrial Fibrillation
Acronym: PVI-PVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tsiachris Dimitrios (Other)
Collaborators: Medtronic Atrial Fibrillation Solutions (Industry)
Responsible Party: Sponsor-Investigator, Tsiachris Dimitrios, Assistant Professor of Cardiology, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4895-18/03/2025
Record Dates: First submitted 2025-06-04; First posted 2025-06-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Catheter Ablation; Pulmonary Vein Isolation
Keywords: Atrial Fibrillation (AF); Pulsed Field Ablation (PFA); Catheter Ablation; Electroanatomical Mapping; Pulmonary Vein Isolation (PVI); Fluoroscopy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoroscopy-based catheter ablation by means of PulseSelect catheter (Device) (Active Comparator): In 20 patients, a fluoroscopy-based approach will be used for visualization of the PulseSelect catheter.
  Interventions: Device: Fluoro based pulmonary vein ablation
- EAM-based catheter ablation by means of PulseSelect catheter (Device) (Active Comparator): In 20 patients Carto 3 Prime® 3D-EAM system (Biosense Webster, Diamond Bar CA) system will be used for visualization of the PulseSelect catheter.
  Initially, a multipolar catheter (PentaRay®) will be used to map the left atrium pre-ablation.
  Interventions: Device: EAM based Pulmonary Vein Isolation

INTERVENTIONS:
Device: EAM based Pulmonary Vein Isolation — 20 patients with symptomatic paroxysmal or persistent AF will be scheduled for pulmonary vein isolation (PVI) based to EAM by means of the PulseSelect catheter.
  Ablation will be performed in a deep sedation setting and additional ablation within the pulmonary veins will be assessed
  Other Names: Catheter Ablation
  Arms: EAM-based catheter ablation by means of PulseSelect catheter (Device)
Device: Fluoro based pulmonary vein ablation — 20 patients with symptomatic paroxysmal or persistent AF will be scheduled for pulmonary vein isolation (PVI) based to Fluoroscopy by means of the PulseSelect catheter.
  Ablation will be performed in a deep sedation setting and additional ablation within the pulmonary veins will be assessed
  Arms: Fluoroscopy-based catheter ablation by means of PulseSelect catheter (Device)

SUMMARY:
Electroanatomical mapping (EAM) based pulmonary vein isolation (PVI) by means of PulseSelect catheter and deep sedation will be compared to fluoroscopy based pulmonary vein isolation in patients with atrial fibrillation in the acute and long term (2 months remapping).

DETAILED DESCRIPTION:
* Trial Population All patients with symptomatic paroxysmal or persistent AF scheduled for PVI
* Treatment Patients with AF will have to receive first oral anticoagulation for 3 weeks. Thereafter all patients will be randomized either to fluoroscopy-based or EAM-based PVI by means of the PulseSelect catheter. Transesophageal echocardiography will not be necessary prior to cardioversion of catheter ablation. Oral anticoagulation will be continued until the morning of the procedure and resumed on the evening after the intervention.
* Deep sedation Patients will be under deep sedation using boluses of midazolam, fentanyl, and propofol. Sedation will be initiated with an intravenous injection of a bolus of 1 to 2 mg midazolam plus 20 to 30 mg propofol. To maintain deep sedation, additional boluses of 10 to 20 mg propofol will be administered at intervals of at least 30 seconds.
* Ablation protocol One application (4 pulse trains) is delivered at each catheter position and a minimum of 8 applications should be completed for each vein, ensuring continuous and overlapping lesions (4 ostial and 4 antral) by rotating the catheter between ablations and flexing the sheath to create overlapping lesion segments. Electrode 5, always distally located, is used as a reference during 45 degrees rotation between each ostial and antral lesion.

EAM use facilitates overlapping and reduces the possibility for gaps. The highlighted fifth electrode is used as quick real-time reference and snapshots of the array immediately prior to pulse delivery as reference for planning subsequent ablation sites.

In both groups an additional set of 4 lesions inside the pulmonary veins will be performed initially before the ostial and antral lesions.

In half patients Carto 3 Prime® 3D-EAM system (Biosense Webster, Diamond Bar CA) system will be used for visualization of the PulseSelect catheter. Initially, a multipolar catheter (PentaRay®) will be used to map the left atrium pre-ablation.

During catheter manipulation, the investigators will visualize both the full array and highlight the fifth electrode to allow for easier and faster perception of the farthest, with regard to catheter shaft, ablation area. Input to the 3D-EAM will be interrupted during energy delivery to prevent malfunction. In cases of an extreme angle of the right inferior pulmonary vein, placement of the PulseSelect catheter in the bottom part of the vein without the guidewire inside the vein may be attempted by means of 3D-EAM and targeting the fifth electrode of the catheter.

The procedural end point will be bidirectional conduction block of all pulmonary veins after a 20-minute observation period. If reconnection of a pulmonary vein is observed, repeat ablation will be performed until block is achieved.

• Follow up/EP Study All patients will be re-assessed 2 months post ablation. Changes of therapy will not be performed during the blind period of 2 months. Clinical atrial tachyarrhythmias recurrence, need for electrical cardioversion and need for hospitalization will also be recorded. A 24-hour holter will be performed 2 months post ablation.

In all patients Carto 3 Prime® 3D-EAM system (Biosense Webster, Diamond Bar CA) system will be used for remapping of the left atrium 2 months post-ablation. All veins will be reassessed for bidirectional block to confirm continued electrical isolation. Any gaps identified will be targeted and ablated with Navistar STSF ablation catheter (Biosense Webster, Diamond Bar CA).

To assess for PV reconnection and the location of gaps, a high-density voltage map will be performed with the color display range set to 0.20 to 0.50 mV as well as to 0.10 to 0.30 mV to accentuate the border zone between healthy tissue and scar for visual identification of gaps. Gaps will be classified according to each PV quarter (anterior, superior, posterior, inferior). Stored fluoroscopy and electroanatomical pamming images from the primary procedure will be used for analysis. In case of PV reconnection, we will search for the earliest activation site as a potential location of a gap. The location of gaps will be defined by PV reisolation during ablation or, in case of multiple gaps, a clear change in PV activation sequence.

In case of aberrant PV anatomy, such as a common left trunk, all PVs were assessed individually for durable isolation and are considered individual PVs in the analyses.

Study follow-up schedule: All patients will be re-assessed at least 2 months post ablation. Changes of therapy will not be performed during the blind period of 2 months. A follow up visit will be performed at least 2 months post ablation. Clinical atrial tachyarrhythmias recurrence, need for electrical cardioversion and need for hospitalization will be recorded. A 24-hour holter will also be performed 2 months post ablation. Likewise, an off-line detailed EAM analysis will be performed post remapping focused on accurate gap identification (if any).

ELIGIBILITY:
Inclusion Criteria:

* ALL the following criteria must be fulfilled:

  1. Male or female patients aged ≥18 and <80 years old.
  2. Patients with paroxysmal or persistent AF requiring PVI.
  3. Signed written informed consent by the patient for participation in the study and agreement to comply with the procedure and the follow-up schedule

Exclusion Criteria:

1. Patients with previous AF ablations
2. EF<35%, CABG surgery within previous 3 months, TIA or stroke within previous 6 months
3. Patients were excluded if ineligible for treatment with oral anticoagulation.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Durability of PVI | 2 to 3 months post index ablation
  Durability of pulmonary vein isolation based on a remap procedure after a follow up of at least 2 months post index procedure (percentage of patients with all PVs isolated, percentage of PVs isolated)
PVI durability by means of a fluoroscopy-based or an EAM-based index procedure | 2 to 3 months post index ablation
  Comparison of PVI durability according to fluoroscopy-based or EAM-based index procedure Number of participants with treatment-related adverse events as assessed by CTCAE v4.0"
Identification of pulmonary vein isolation gaps acutely based on EAM | 2 to 3 months post index ablation
  Mapping will be performed in all cases post PVI (either fluoroscopy-based or EAM-based)
Identification of pulmonary vein isolation gaps on remap | 2 to 3 months post index ablation
  Remapping will be performed 2+ months post-index procedure

SECONDARY OUTCOMES:
Fluoroscopy time and dose | During index procedure
  Fluoroscopy time and dose of the index procedure
First pass pulmonary vein isolation | Index procedure
  Frequency of touch-up applications being required acutely post pulmonary vein isolation
Durability of superior vena cava isolation | 2-3 months post index procedure
  Durability of superior vena cava isolation performed during the index procedure
Procedure time | During index procedure
  Procedure time of the index procedure.
Left atrial access time to sheath removal | During index procedure
  Left atrial access time to sheath removal
Left atrial dwelling time | During index procedure
  Left atrial access time

OTHER OUTCOMES:
Patient Safety | 2-3 months
  * Safety of PFA lesions inside the pulmonary veins in the 2 months remap (pulmonary vein stenosis)
  * Major acute complications of deep sedation and propofol use (need for anesthesiologist, need for intubation, need for ICU hospitalization)
  * Major acute complications of ablation (death, cardiac tamponade not related to transeptal). [Time Frame: Acute peri-procedural complications will be defined as occurring within 24 hours of ablation]

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Cardiology, National and Kapodistrian University of Athens, Hippokration General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kordalis A, Tsiachris D, Antoniou CK, Doundoulakis I, Tsioufis K. Verification of persistent pulmonary vein isolation with electroanatomical mapping 3 months after ablation using a novel PFA platform. Hellenic J Cardiol. 2024 Nov 19:S1109-9666(24)00232-X. doi: 10.1016/j.hjc.2024.11.002. Online ahead of print. No abstract available. PMID 39566605
- [Result] Tsiachris D, Antoniou CK, Doundoulakis I, Kordalis A, Stefanadis C, Tsioufis K. Single-center initial experience with a new pulsed-field ablation system: pulmonary vein isolation lesions and beyond. Future Cardiol. 2024;20(14):739-746. doi: 10.1080/14796678.2024.2413829. Epub 2024 Nov 19. PMID 39560013